CLINICAL TRIAL: NCT04960761
Title: The Effect of Education Given to Children With Audio and Picture Books on Anxiety, Quality of Life and Early Mobilization in the Preoperative Period
Brief Title: The Effectiveness of the Training Given With Audio and Picture Book Before the Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, RN, PhD, Asst Prof. Surgical Nursing, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-21/15
Record Dates: First submitted 2021-06-22; First posted 2021-07-14 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Pediatric ALL; Appendix Diseases
Keywords: anxiety; surgery; child; mobilization; quality of life
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Pre-operative training will be given by the clinic nurse with audio and picture book. Training content with audio and picture book; Before the operation, the procedures performed during the admission of the patient to the service (introducing the clinic and staff to the patient), what are the preoperative preparations (checking vital signs, intravenous (IV) catheter application, wearing a surgical gown), wearing a patient tag on the wrist, taking him to the operating room on a stretcher), which will be used during the operation anesthesia techniques and how to provide sedation (the anesthetic agent can be given by mask or IV catheter, the reasons are the clothes worn by doctors and nurses in the operating room), what are the procedures that can be applied after the surgery (vital signs control, monitoring, oxygen administration, serum insertion, etc.).
  Interventions: Other: İntervention Group
- Control Group (No Intervention): Routine training will be given by a nurse working in the clinic during the preoperative period. The content of the routine training: What are the procedures performed during the admission of the patient to the service before the operation (introducing the clinic and the staff to the patient), what the preoperative preparation is (checking vital signs, intravenous (IV) catheter application, wearing a surgical gown, wearing a patient tag on the wrist, with a stretcher. being taken to the operating room), what are the procedures that can be applied after the surgery (vital signs control, monitoring, oxygen administration, serum insertion, etc.), there may be some medical materials that were applied to the patient during the surgery (nasogastric tube, IV catheter, types of drains placed in the wound site) includes information such as

INTERVENTIONS:
Other: İntervention Group — In the experimental group, pre-operative anxiety and quality of life scales will be applied to the child and their parents before and after the operation with audio and picture books, the preoperative quality of life scale will be made, the postoperative anxiety and quality of life scale will be repeated and the early mobilization scale will be made.
  The control group will be routinely informed before the operation, an anxiety scale will be given to the child and their parents before the operation, a quality of life scale will be given to the child, the postoperative anxiety and quality of life scale will be repeated, and early mobilization form will be applied.
  Other Names: Control Group
  Arms: Intervention Group

SUMMARY:
Behavioral practices applied to the child in the preoperative period; It includes methods such as introducing the hospital and operating room to children and their parents, reading storybooks, giving training books, an educational internet application with interactive games, and using visual aids. At the same time, by using an appropriate anatomy book, it can help the child to visualize his body correctly, to understand the size and location of the surgical site, and to learn where the suture will be after the intervention.In this study, it was aimed to evaluate the effect of preoperative education with the help of audio and picture books on postoperative anxiety, quality of life and early mobilization.

DETAILED DESCRIPTION:
Psychological preparation process in the pre-operative period; It reduces anxiety, uses less anesthetic during the operation, normalizes vital signs in a short time, uses less painkillers and helps early discharge. Behavioral practices applied to the child in the preoperative period; It includes methods such as introducing the hospital and operating room to children and their parents, reading storybooks, giving training booklets, an educational internet application with interactive games, and using visual aids. At the same time, by using an appropriate anatomy book, it can help the child to visualize his body correctly, to understand the size and location of the surgical site, and to learn where the suture will be after the intervention. No study was found in which children aged 8-12 years were educated with the help of audio and picture books before appendectomy and evaluated postoperative anxiety, quality of life and mobilization time. In this study, it was aimed to evaluate the effect of preoperative education with the help of audio and picture books on postoperative anxiety, quality of life and early mobilization. The study was planned randomized controlled study. The statistical universe of this study, includes pediatric patients who operated between February 2021 and December 2021 in Pediatric Surgery Department in Zeynep Kamil Maternity and Children's hospital. The sample includes who operated with appendectomy between the ages of 8 and 12 who met the inclusion criteria in the Pediatric Surgery Clinic as 60 children. Participants will be divided into two equal groups as intervention (n=30) and control (n=30) groups. Children and Parents Descriptive Characteristics Form, State Anxiety Inventory for Children, State Anxiety Inventory (for Parents), Quality of Life Scale for Children, Evaluation of Postoperative Mobilization Time will be used to collect data. Data will be analyzed with appropriate statistical methods using the SPSS for Windows 22.0 program (Statistical Package for the Social Sciences). Descriptive statistical methods such as percentile, mean, standard deviation and median in the evaluation of data and Kolmogorov-Smirnov distribution test for examining normal distribution, chi-square test, t-test/Mann Whitney-U test for measurement data, One-Way ANOVA/Kruskall Wallis tests will be used.

ELIGIBILITY:
Inclusion Criteria:

* Child criteria

  * Be between 8-12 years old
  * Having an appendectomy operation
  * ASA classification I and II
  * Staying in hospital for at least 24 hours after surgery
* Parent criteria

  * Being literate
  * The child's mother or father
  * Parent can use smartphone

Exclusion Criteria:

* Parent/child not accepting the research
* Presence of a parent/child's mental disability

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-08-31 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Determining the change in children's anxiety levels with the state anxiety inventory for children | Preoperative period(one hour before surgery) and one day after surgery
  The measure of this study is to determine the effect of informing with audio and picture books on children's anxiety in the preoperative period with the state anxiety inventory for children.
Determination of the change in parents' anxiety levels with the state anxiety inventory for parents | Preoperative period(one hour before surgery) and one day after surgery
  The measure of this study is to determine the effect of parental state anxiety inventory and preoperative information with audio and picture books on parents' anxiety.

SECONDARY OUTCOMES:
Determination of the change in quality of life levels of children with the quality of life scale for children | Preoperative period(one hour before surgery) and one day after surgery
  The measure of this study is to determine the change in quality life of children, who are informed with audio and picture books before surgery, and the effectiveness with the quality of life scale for children.
Determination of the change in the mobilization time of children after the surgery with the mobilization time form for children | About 4-6 hours after surgery
  The measure of this study is to determine the change in mobilization time of children, who are informed with audio and picture books before surgery, with the mobilization form.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ono S, Oikawa I, Hirabayashi Y, Manabe Y. Preparation of a picture book to support parents and autonomy in preschool children facing day surgery. Pediatr Nurs. 2008 Jan-Feb;34(1):82-3, 88. No abstract available. PMID 18361093
- [Background] Nilsson E, Svensson G, Frisman GH. Picture book support for preparing children ahead of and during day surgery. Nurs Child Young People. 2016 Oct 7;28(8):30-35. doi: 10.7748/ncyp.2016.e749. PMID 27712311
- [Background] Kain ZN, Caramico LA, Mayes LC, Genevro JL, Bornstein MH, Hofstadter MB. Preoperative preparation programs in children: a comparative examination. Anesth Analg. 1998 Dec;87(6):1249-55. doi: 10.1097/00000539-199812000-00007. PMID 9842807
- [Background] Coskunturk AE, Gozen D. The Effect of Interactive Therapeutic Play Education Program on Anxiety Levels of Children Undergoing Cardiac Surgery and Their Mothers. J Perianesth Nurs. 2018 Dec;33(6):781-789. doi: 10.1016/j.jopan.2017.07.009. Epub 2018 Feb 3. PMID 29398304
- [Background] Hatava P, Olsson GL, Lagerkranser M. Preoperative psychological preparation for children undergoing ENT operations: a comparison of two methods. Paediatr Anaesth. 2000;10(5):477-86. doi: 10.1046/j.1460-9592.2000.00537.x. PMID 11012950
- [Background] Li HC, Lopez V. Effectiveness and appropriateness of therapeutic play intervention in preparing children for surgery: a randomized controlled trial study. J Spec Pediatr Nurs. 2008 Apr;13(2):63-73. doi: 10.1111/j.1744-6155.2008.00138.x. PMID 18366374